CLINICAL TRIAL: NCT03613129
Title: Pilot Phase 1/2, Open-Label, Clinical Trial to Investigate CT38 in the Treatment of Myalgic Encephalomyelitis / Chronic Fatigue Syndrome
Brief Title: Clinical Trial to Investigate CT38 in the Treatment of Myalgic Encephalomyelitis / Chronic Fatigue Syndrome
Acronym: InTiME
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LUCINDA BATEMAN, MD (Other)
Responsible Party: Sponsor-Investigator, LUCINDA BATEMAN, MD, Founder & Medical Director, Bateman Horne Center
Organization: Bateman Horne Center (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ME-101p
Record Dates: First submitted 2018-07-13; First posted 2018-08-02 (Actual); Results first posted 2020-04-30 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Myalgic Encephalomyelitis; Chronic Fatigue Syndrome
Keywords: myalgic encephalomyelitis; chronic fatigue syndrome; corticotropin releasing-factor receptor subtype 2 (CRF2); Alternative CRF2 names: CRFR2, CRH2, CRHR2
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Intervention Model Description: The study is comprised of a recruitment and screening period, enrollment (Visit 1), a 4-week (at least) pre-treatment assessment period, a 1-week interventional treatment period with drug infused at Visits 3, 4 and 4b, a 4-week (at least) post-treatment assessment period, and a close-out (Visit 6).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- D0.20 (Active Comparator): Subcutaneous infusion of CT38 at 0.20 μg/kg/hour, for 3 hours on each of 2 days
  Interventions: Drug: CT38
- D0.03 (Active Comparator): Subcutaneous infusion of CT38 at 0.03 μg/kg/hour, for 3.5 hours on each of 3 days
  Interventions: Drug: CT38
- D0.06 (Active Comparator): Subcutaneous infusion of CT38 at 0.06 μg/kg/hour, for 3.5 hours on each of 3 days
  Interventions: Drug: CT38
- D0.01 (Active Comparator): Subcutaneous infusion of CT38 at 0.01 μg/kg/hour, for 3.5 hours on each of 3 days
  Interventions: Drug: CT38

INTERVENTIONS:
Drug: CT38 — Infusion

SUMMARY:
This study seeks to investigate the safety, tolerability and efficacy of CT38, an experimental peptide administered by subcutaneous infusion, in the treatment of ME/CFS patients.

DETAILED DESCRIPTION:
Myalgic Encephalomyelitis / Chronic Fatigue Syndrome (ME/CFS) is a complex disorder that may be triggered by infection or other stressors (e.g., emotional or physical trauma, immune activation, chemical exposures). Its hallmark is a reduced capacity for physical and mental activity manifest as profound fatigue along with a cascade of debilitating symptoms (including pain, cognitive dysfunction, orthostatic intolerance, sensitivities, and irregularities of the autonomic, immune and metabolic systems) that worsen with activity (referred to as post-exertional malaise or PEM), are not improved by sleep, and can persist for years. Patients are often unable to handle the activities of daily living and experience a loss of career and a very poor quality of life. There are no established diagnostic tests or approved therapeutics for ME/CFS.

The cause of ME/CFS is not known. It has been postulated that ME/CFS could arise from the up-regulation of a specific receptor (CRF2) in those parts of the brain that govern the sensitivity of the stress response. This configuration would invoke a major response to a minor stimulus, ultimately leading to neuroendocrine, autonomic, immune and metabolic abnormalities that are commonly observed. There is no animal model of ME/CFS, but overstimulating CRF2 in healthy rats, induces signs and symptoms consistent with the disease in humans; while down-regulating it, via CT38 (an experimental peptide), eliminates the ability to stimulate these signs and symptoms. Hypothesis: Utilize CT38 to down-regulate CRF2 to restore a normal stress response, and potentially eliminate disease signs and symptoms.

The study will enroll 18 patients, who meet the Fukuda and Canadian criteria for ME/CFS, and treat them with various doses of CT38.

The primary endpoint will be the change in the average total daily symptom score (TDSS), over 28-day periods immediately prior to the first treatment (pre-treatment) and immediately prior to exit from the trial (post-treatment). The TDSS is the sum of 13 individual symptom scores, each recorded daily by the patient on a 6-point scale (0=none, 1=very mild, 2=mild, 3=moderate, 4=severe, 5=very severe). The individual symptoms included fatigue, muscle/joint pain, sleep issues (e.g., un-refreshing sleep, difficulty falling or staying asleep, excessive sleepiness), cognitive issues (e.g., slow information processing, memory difficulties, inability to concentrate/focus, attention deficit), orthostatic intolerance (e.g., dizziness, spatial disorientation, light-headedness, feeling faint), body temperature perceptions, flu-like symptoms (e.g., sore throat, tender lymph nodes, swollen glands, fever, chills, sinus/nasal problems), headaches or sensory sensitivities (to light, sound, smell, touch, taste), shortness of breath, gastrointestinal problems (e.g., nausea, stomach/abdominal pain, diarrhea), urogenital problems (e.g., frequent urination), anxiety and depression.

The secondary outcomes will assess general health status (determined by Short-Form 36, or SF-36), as well as safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Ability to read, understand and speak English
* Living at an altitude between 3,500 and 5,500 feet above sea level for the past 1 year
* Willing to perform an exercise test
* Diagnosed with ME/CFS and meet the following 3 case definitions: Fukuda Research Case Definition for CFS (1994), Revised Canadian Consensus Criteria for ME/CFS (2010) and the Institute of Medicine (IOM) Clinical Diagnostic Criteria for ME/CFS (2015)
* Relatively stable state of illness for the individual patient over the past 3 months
* Male or female, between the ages of 18 and 60 years old
* Males or females of reproductive potential agree to remain abstinent or use (or have their partner use) 2 acceptable methods of contraception, starting from the time of informed consent through 28 days after the last dose of study drug. Acceptable methods of birth control during the study are intrauterine device, diaphragm with spermicide, contraceptive sponge, condom or vasectomy. Oral contraceptive pills may not be used as the sole method of contraception because the effect of CT38 on the efficacy of oral contraceptive pills has not yet been established
* Stated willingness to comply with all study procedures and remain available for the study duration
* Have mobile (smart) phone and access to the internet

Exclusion Criteria:

* Alternate medical or psychiatric illness that could explain the ME/CFS symptoms
* Unwilling or unable to perform an exercise test
* Active or uncontrolled co-morbidities which in the opinion of the PI may interfere with the ability of the patient to participate in the study. Co-morbidities may include acute infection, Crohn's disease, diabetes mellitus (Type 1 or Type 2, evidenced by a history of glycated hemoglobin (A1C) > 7 at any time), Guillain-Barre syndrome, lupus, multiple sclerosis, myasthenia gravis, rheumatoid arthritis, or other such diseases that may be exclusionary. Particularly conditions or medications that cause immunodeficiency or immunosuppression will be excluded. Examples of such conditions can be found in the tables "Causes of Secondary Immunodeficiency" and "Some Drugs that Cause Immunosuppression" in the "Merck Manual"
* Pregnancy, or while breast feeding. Women should not be enrolled within 6 months of giving birth and within 3 months of cessation of breast feeding
* A Body Mass Index > 35
* Cigarette smoker or former smoker who has smoked within 6 months of the start of the study
* Living at an altitude that is more than 1,000 feet (lower or higher) from the study site (which is 4,500 feet above sea level)
* History of:

  * Major depression with psychotic or melancholic features before the diagnosis of ME/CFS, or active depression (major depression with psychotic or melancholic features) as determined by self-report
  * Untreated endocrine diagnoses including hypothyroidism (Hashimoto's, etc.), Grave's disease, adrenal insufficiency, hypogonadism (testosterone deficiency), diabetes mellitus or insipidus
  * Acute infection within the past 30 days
  * Within the last 3 years, any significant head injury, e.g., concussion with loss of consciousness, brain surgery, an automobile accident with head/neck injury, other traumatic brain injury
  * A supra-ventricular tachycardia or ventricular tachycardia, e.g., atrial fibrillation or flutter, paroxysmal atrial fibrillation, junctional tachycardia, ventricular tachycardia
  * Severe baseline hypotension defined as rested sitting systolic BP < 100 mmHg or rested sitting diastolic BP < 60 mmHg
  * Renal impairment based upon the local lab normal estimated glomerular filtration rate (eGFR) (drug is cleared by passive renal filtration)
  * Known hypersensitivity or clinically significant allergies to tromethamine or Tween 80 (both excipients in the drug product)
  * Substance abuse in the past 12 months as determined by self-report
* Improvement in overall ME/CFS symptoms as a result of any treatment intervention in the past 3 months
* Current treatment with medications that interact with pathways involving: (i) 5-hydroxytryptamine (5HT) (e.g., selective 5HT re-uptake inhibitors or selective serotonin reuptake inhibitors (SSRIs), 5HT and norepinephrine re-uptake inhibitors or serotonin and norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, monoamine oxidase inhibitors, triptans); (ii) norepinephrine (e.g., adrenergic agonists or antagonists, norepinephrine re-uptake inhibitors, norepinephrine and dopamine re- uptake inhibitors); (iii) dopamine (e.g., norepinephrine and dopamine re-uptake inhibitors); and (iv) cortisol pathways (e.g., oral glucocorticoids, fludrocortisone).
* Prior treatment with

  * Short-term (< 2 weeks) antiviral or antibiotic medication or flu shot within the past 4 weeks
  * Long-term (> 2 weeks) antiretrovirals within the past 12 months
  * RituximabTM within 6 months
  * Any new prescription drug or herbal remedy within 2 weeks prior to the onset of the trial
* Current participation in another clinical treatment trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucinda Bateman, MD, Principal Investigator — Bateman Horne Center; Suzanne D Vernon, PhD, Study Director — Bateman Horne Center
Locations (1):
- Bateman Horne Center, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Pereira G, Gillies H, Chanda S, Corbett M, Vernon SD, Milani T, Bateman L. Acute Corticotropin-Releasing Factor Receptor Type 2 Agonism Results in Sustained Symptom Improvement in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome. Front Syst Neurosci. 2021 Sep 1;15:698240. doi: 10.3389/fnsys.2021.698240. eCollection 2021. PMID 34539356

RESULTS

PARTICIPANT FLOW:
Groups:
- Screen Failures: Patient enrolled, but screened-out before receiving treatment
Period: Pre-treatment Assessment
Arm/Group | Screen Failures | D0.01 | D0.03 | D0.06 | D0.20
Started | 3 | 3 | 7 | 2 | 2
Completed | 0 | 3 | 7 | 2 | 2
Not Completed | 3 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Period: Treatment
Arm/Group | Screen Failures | D0.01 | D0.03 | D0.06 | D0.20
Started | 0 | 3 | 7 | 2 | 2
Completed | 0 | 3 (ID35 received only 1 infusion (due to symptom worsening)) | 7 | 2 (ID34 did not receive 3rd infusion (for lack of venous access)) | 2
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Post-treatment Assessment
Arm/Group | Screen Failures | D0.01 | D0.03 | D0.06 | D0.20
Started | 0 | 3 | 7 | 2 | 2
Completed | 0 | 3 | 7 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D0.01 | D0.03 | D0.06 | D0.20 | Total
Number analyzed (Participants) | 3 | 7 | 2 | 2 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (8.2) | 39.7 (7.2) | 53.6 (0.6) | 44.6 (21.4) | 43.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 2 | 0 | 8
  Male | 2 | 2 | 0 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 5 | 2 | 2 | 12
  Other | 0 | 2 | 0 | 0 | 2
Age, at diagnosis [Mean (Standard Deviation); unit: years] | 33.7 (12.2) | 32.4 (10.4) | 46.0 (9.9) | 32.5 (24.7) | 34.6 (12.3)
Disease onset [Count of Participants; unit: Participants]
  Gradual | 2 | 3 | 1 | 2 | 8
  Sudden | 1 | 4 | 1 | 0 | 6
Disease triggers [Count of Participants; unit: Participants]
  Infection | 3 | 6 | 2 | 2 | 13
  Toxins | 1 | 2 | 0 | 1 | 4
  Over-exertion | 0 | 1 | 1 | 0 | 2
  Emotion | 0 | 3 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Total Daily Symptom Score (TDSS)
Description: Pre-/post-treatment difference in TDSS (0-65 scale, 0=no symptoms; 65=maximum of 5 for each of 13 specific patient-reported symptoms). The TDSS sums the patient-reported daily symptom score for each of 13 specific symptoms (including fatigue, muscle/joint pain, sleep problems, cognitive problems, orthostatic intolerance, body temperature perceptions, flu-like symptoms, headaches or sensitivities, shortness of breath, gastrointestinal problems, urogenital problems, anxiety and depression), each assessed on a 0-5 scale (0=no symptom, 1=very mild, 2=mild, 3=moderate, 4=severe, 5=severe)
Time Frame: 28 days preceding Visit 3 (pre-treatment) and 28 days preceding Visit 6 (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intent-to-treat: All patients receiving test drug
Arm/Group | Intent-to-treat | D0.01 | D0.03 | D0.06 | D0.20
Number analyzed (Participants) | 14 | 3 | 7 | 2 | 2
units on a scale
  Pre-treatment TDSS | 29.5 (9.4) | 28.7 (12.2) | 29.2 (11.4) | 31.3 (1.3) | 30.1 (8.0)
  Post-treatment TDSS | 25.3 (9.6) | 25.5 (10.5) | 21.7 (10.3) | 29.5 (3.5) | 33.0 (9.6)
Statistical Analysis 1: Comparison: Intent-to-treat; Test type: Non-Inferiority — Comparing 28-day pre-treatment mean TDSS and 28-day post-treatment mean TDSS; p = 0.011, t-test, 2 sided
Statistical Analysis 2: Comparison: D0.01; Test type: Non-Inferiority — Comparing 28-day pre-treatment mean TDSS and 28-day post-treatment mean TDSS; p = 0.136, t-test, 2 sided
Statistical Analysis 3: Comparison: D0.03; Test type: Non-Inferiority — Comparing 28-day pre-treatment mean TDSS and 28-day post-treatment mean TDSS; p = 0.009, t-test, 2 sided
Statistical Analysis 4: Comparison: D0.06; Test type: Non-Inferiority — Comparing 28-day pre-treatment mean TDSS and 28-day post-treatment mean TDSS; p = 0.451, t-test, 2 sided
Statistical Analysis 5: Comparison: D0.20; Test type: Non-Inferiority — Comparing 28-day pre-treatment mean TDSS and 28-day post-treatment mean TDSS; p = 0.240, t-test, 2 sided

2. Secondary Outcome: SF-36, PCS
Description: Pre-/post-treatment difference in the physical component score (PCS) of the RAND 36-Item Health Survey (SF-36), on a 0-100 scale (where 0=max disability and 100=no disability)
Time Frame: Visit 3 before treatment (pre-treatment) and at Visit 6 (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intent-to-treat | D0.01 | D0.03 | D0.06 | D0.20
Number analyzed (Participants) | 14 | 3 | 7 | 2 | 2
units on a scale
  Pre-treatment PCS | 27.9 (4.0) | 25.9 (6.9) | 24.6 (3.7) | 27.6 (1.4) | 30.6 (1.4)
  Post-treatment PCS | 31.5 (5.8) | 29.1 (6.0) | 30.7 (5.3) | 27.0 (1.4) | 26.8 (0.9)
Statistical Analysis 1: Comparison: Intent-to-treat; Test type: Non-Inferiority — Comparing pre-treatment PCS (at Visit 3) and post-treatment PCS (at Visit 6); p = 0.039, t-test, 2 sided
Statistical Analysis 2: Comparison: D0.01; Test type: Non-Inferiority — Comparing pre-treatment PCS (at Visit 3) and post-treatment PCS (at Visit 6); p = 0.191, t-test, 2 sided
Statistical Analysis 3: Comparison: D0.03; Test type: Non-Inferiority — Comparing pre-treatment PCS (at Visit 3) and post-treatment PCS (at Visit 6); p = 0.016, t-test, 2 sided
Statistical Analysis 4: Comparison: D0.06; Test type: Non-Inferiority — Comparing pre-treatment PCS (at Visit 3) and post-treatment PCS (at Visit 6); p = 0.053, t-test, 2 sided
Statistical Analysis 5: Comparison: D0.20; Test type: Non-Inferiority — Comparing pre-treatment PCS (at Visit 3) and post-treatment PCS (at Visit 6); p = 0.060, t-test, 2 sided

3. Secondary Outcome: SF-36, MCS
Description: Pre-/post-treatment difference in the mental component score (MCS) of the RAND 36-Item Health Survey (SF-36), on a 0-100 scale (where 0=max disability and 100=no disability)
Time Frame: Visit 3 before treatment (pre-treatment) and at Visit 6 (post-treatment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intent-to-treat | D0.01 | D0.03 | D0.06 | D0.20
Number analyzed (Participants) | 14 | 3 | 7 | 2 | 2
units on a scale
  Pre-treatment MCS | 34.0 (3.6) | 36.3 (3.2) | 28.9 (3.9) | 32.1 (3.2) | 35.8 (2.6)
  Post-treatment MCS | 34.8 (6.3) | 38.5 (9.1) | 29.9 (6.4) | 34.9 (5.6) | 31.5 (2.1)
Statistical Analysis 1: Comparison: Intent-to-treat; Test type: Non-Inferiority — Comparing pre-treatment MCS (at Visit 3) and post-treatment MCS (at Visit 6); p = 0.587, t-test, 2 sided
Statistical Analysis 2: Comparison: D0.01; Test type: Non-Inferiority — Comparing pre-treatment MCS (at Visit 3) and post-treatment MCS (at Visit 6); p = 0.618, t-test, 2 sided
Statistical Analysis 3: Comparison: D0.03; Test type: Non-Inferiority — Comparing pre-treatment MCS (at Visit 3) and post-treatment MCS (at Visit 6); p = 0.634, t-test, 2 sided
Statistical Analysis 4: Comparison: D0.06; Test type: Non-Inferiority — Comparing pre-treatment MCS (at Visit 3) and post-treatment MCS (at Visit 6); p = 0.355, t-test, 2 sided
Statistical Analysis 5: Comparison: D0.20; Test type: Non-Inferiority — Comparing pre-treatment MCS (at Visit 3) and post-treatment MCS (at Visit 6); p = 0.417, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: At least 10 weeks
Arm/Group | Intent-to-treat | D0.01 | D0.03 | D0.06 | D0.20
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/3 | 0/7 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/3 | 0/7 | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 14/14 | 3/3 | 7/7 | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-treat (N=14) | D0.01 (N=3) | D0.03 (N=7) | D0.06 (N=2) | D0.20 (N=2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Tachycardia resulting from too high a first-in-patient dose (predicted from healthy animals/humans that could not account for CRF2 upregulation), and an inadvertent protocol deviation that continued dosing after the dose-stopping criteria were met
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hypotension resulting from too high a first-in-patient dose (predicted from healthy animals/humans that could not account for CRF2 upregulation), and an inadvertent protocol deviation that continued dosing after the dose-stopping criteria were met
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intent-to-treat (N=14) | D0.01 (N=3) | D0.03 (N=7) | D0.06 (N=2) | D0.20 (N=2)
Swollen lymph nodes (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (5) | 0 (0) | 1 (3) | 1 (2) | 0 (0)
Premature ventricular contraction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperemic eyes (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Sore throat (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Body aches (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature abnormalities (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (10) | 0 (0) | 3 (5) | 0 (0) | 2 (5)
Influenza like illness (General disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Myalgia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain & discomfort (General disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (Musculoskeletal and connective tissue disorders) | 3 (6) | 1 (4) | 1 (1) | 0 (0) | 1 (1)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Forgetfulness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (18) | 3 (6) | 5 (8) | 2 (3) | 1 (1)
Restlessness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wired (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysequilibrium (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Anxiety State (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disturbance (Psychiatric disorders) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Emotional lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder disturbance (Psychiatric disorders) | 6 (7) | 1 (1) | 4 (5) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sinus infection (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Facial flushing (Vascular disorders) | 6 (10) | 1 (1) | 3 (7) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 13 (27) | 3 (6) | 6 (14) | 2 (5) | 2 (2)
Hot flushes (Vascular disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pallor (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
InTiME was based on a novel theory of ME/CFS and an unprecedented drug mechanism. Predicted doses had to be adjusted, limiting statistical inferences, but providing preliminary support for the hypothesis and treatment approach.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT03613129/Prot_SAP_000.pdf